CLINICAL TRIAL: NCT05974527
Title: Pilot Study 1: Efficacy and Safety of Sublingual Dexmedetomidine (BXCL501) for the Treatment of Agitation in the Emergency Department
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study did not start - due to funding issues prior to IRB approval
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Dana Im, MD, MPHIL, MPP, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023p001864
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Agitation; Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders; Bipolar Disorder
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention - BXCL501 (Experimental)
  Interventions: Drug: Sublingual film containing dexmedetomidine (BXCL501)

INTERVENTIONS:
Drug: Sublingual film containing dexmedetomidine (BXCL501) — Enrolled participants will receive an initial dose of BXCL501 180mcg. Following the FDA dosing suggestions, participants with mild or moderate hepatic impairment (Child-Pugh Class A or B) will receive a reduced initial dose of 120mcg and participants with severe hepatic impairment (Child-Pugh Class C) will receive a reduced initial dose of 90mcg. Geriatric patients (≥ 65 years old) will receive a reduced initial dose of 120mcg.

SUMMARY:
This is a single-arm pilot study to examine the impact of BXCL501 (sublingual film formulation of dexmedetomidine) administration on reducing the severity of undifferentiated acute agitation in patients presenting to the emergency department with underlying bipolar disorder or schizophrenia. This study is designed to evaluate BXCL501 for its FDA-approved indication -- treatment of agitation associated with bipolar disorder or schizophrenia -- applied in the emergency department setting.

DETAILED DESCRIPTION:
This pilot study will enroll 30 male and female adults with primary psychiatric complaint and a documented diagnosis of bipolar I disorder, bipolar II disorder, schizophrenia, schizoaffective disorder, or schizophreniform disorder, presenting to the emergency department with clinical signs of acute agitation. Eligible subjects will receive an initial dose of BXCL501 (180mcg) and a repeat dose (90mcg) 2 hours after the first BXCL501 dose in the event of persistent or recurrent agitation (up to two repeat doses) while under medical supervision in the emergency department. Efficacy and safety assessments will be conducted periodically before and after dosing.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults age ≥18 years
* Patients with an established diagnosis of (1) bipolar I disorder, (2) bipolar II disorder, (3) schizophrenia, (4) schizoaffective disorder, or (5) schizophreniform disorder
* Judged to be clinically agitated at the time of Screening and Baseline with a AMSS ≥2
* Able to read, understand, and provide written informed consent
* Subject judged to be likely capable of self-administration of BXCL501 sublingually or buccally

Exclusion Criteria:

* Likely to be discharged, admitted, or transferred from the ED within 6 hours after study medication administration
* Administration of benzodiazepines or antipsychotic drugs in the 2 hours before study treatment
* Treatment with alpha-1 noradrenergic antagonists
* Female patients who are pregnant or are breastfeeding
* Hypotension (systolic blood pressure <100 mmHg or diastolic blood pressure <60 mmHg) and/or bradycardia (heart rate <55 beats per minute) at the time of Screening or Baseline evaluation
* History of dysautonomia
* Patient with a known diagnosis of familial long QT syndrome, second degree or third degree atrioventricular block without pacemaker, or sick sinus syndrome
* Patients with serious or unstable medical illnesses determined by the study investigators or qualified designees
* Patients with history of allergic reactions to dexmedetomidine
* Patients previously enrolled and completed the current study
* Patients actively enrolled in other ED-based studies involving pharmacological or behavioral interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in the Altered Mental Status Scale (AMSS) score | 120 minutes
  AMSS is a 9-point scale ranging from -4 (most sedated) to 4 (most agitated).

SECONDARY OUTCOMES:
Absolute change from baseline in the Richmond Agitation Sedation Scale (RASS) score | 120 minutes
  RASS is a 10-point scale with four levels of anxiety or agitation (+1 to +4), one denoting a calm, alert state (0), and five levels of sedation (-1 to -5).
Absolute change from baseline in the Behavioral Activity Rating Scale (BARS) score | 120 minutes
  BARS is a 7-point scale ranging from 1 (difficult or unable to arouse) to 7 (violent, requires restraints).
Absolute change from baseline in the Broset Violence Checklist (BVC) score | 120 minutes
  BVC is a six-item instrument with a total score ranging from 0 (no agitation) to 6 (severely agitated).
Times, in minutes, from BXCL501 administration to adequate sedation, defined as Altered Mental Status Scale (AMSS) score <1 | To be determined - will be measured for 120 minutes
  AMSS is a 9-point scale ranging from -4 (most sedated) to 4 (most agitated).
Times, in minutes, from BXCL501 administration to adequate sedation, defined as Richmond Agitation Sedation Scale (RASS) score <1 | To be determined - will be measured for 120 minutes
  RASS is a 10-point scale with four levels of anxiety or agitation (+1 to +4), one denoting a calm, alert state (0), and five levels of sedation (-1 to -5).
Times, in minutes, from BXCL501 administration to adequate sedation, defined as Behavioral Activity Rating Scale (BARS) score <5 | To be determined - will be measured for 120 minutes
  BARS is a 7-point scale ranging from 1 (difficult or unable to arouse) to 7 (violent, requires restraints).
Times, in minutes, from BXCL501 administration to adequate sedation, defined as Broset Violence Checklist (BVC) score <1 | To be determined - will be measured for 120 minutes
  BVC is a six-item instrument with a total score ranging from 0 (no agitation) to 6 (severely agitated).